CLINICAL TRIAL: NCT04374006
Title: Effects of Tetragonula Aff. Biroi Propolis Extract on Lesion Growth, Apoptotic and Inflammatory Activity of the Rat Endometriosis Tissue
Brief Title: Effects of Sulawesi Propolis Extract on Lesion Growth, Apoptotic and Inflammatory Activity of the Rat Endometriosis Tissue
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr Herbert Situmorang,SpOG(K), Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-10-1269'
Record Dates: First submitted 2020-04-21; First posted 2020-05-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Endometriosis; Peritoneum; Endometriosis
Keywords: endometriosis; propolis
MeSH Terms: conditions — Endometriosis | interventions — dienogest; Propolis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- propolis 50 (Experimental): we do sonde everyday to the rat that given treatment of 50mg/kg propolis for 2, 4, and 6 weeks
  Interventions: Drug: Propolis
- propolis 100 (Experimental): we do sonde everyday to the rat that given treatment of 100mg/kg propolis for 2, 4, and 6 weeks
  Interventions: Drug: Propolis
- dienogest (Active Comparator): we do sonde everyday to the rat that given treatment of 25mg/kg dienogest for 2, 4, and 6 weeks
  Interventions: Drug: Dienogest
- water (Placebo Comparator): we do sonde everyday to the rat that given 0,2 ml water placebo for 2, 4, and 6 weeks
  Interventions: Other: placebo
- sham group (Sham Comparator): after the 2nd laparotomy, we do nothing about sonde, just giving food and drink everyday
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Dienogest — 1mg/kg BW/day based on the study by Katayama et al. A DNG in 0,5% carboxymethylcellulose suspension was given orally with metal sound daily 0,2-0,4 mL per day
  Other Names: visanne
  Arms: dienogest
Drug: Propolis — The propolis contains 20 mg in each ml. So, each rat we given 0,2 ml for 50mg/kg propolis treatment and 0,4 ml for 100mg/kg propolis treatment
  Other Names: sulawesian propolis
  Arms: propolis 100; propolis 50
Other: placebo — we gave 0,2 ml to each rat everyday to negative control groups, and we gave no treatment to sham groups
  Arms: sham group; water

SUMMARY:
This study aims to evaluating inflammatory and apoptotic activity in rat's endometriosis lesion treated by Propolis compared to Dienogest

DETAILED DESCRIPTION:
Propolis has known of having various efficacy. The main benefits are as antimicrobial, antioxidant, anti-inflammatory, immunomodulatory and antiapoptotic.Propolis has even been shown to have an antibacterial effect in vitro, without requiring human immunological reactions.

The immunological effect of propolis is generated through immune suppression directly and decreasing cytokine production which stimulates immune process. Although proven to have a various efficacy, propolis can't be used as a therapeutic drug due to the difficulty of obtaining standard chemical composition as a requirement to be the drug's substances. Therefore, it is necessary to have biological composition in each propolis prepartions written down before comparing the efficacy.

Anti tumor activity by propolis, which has been tested in animal previously, showed that propolis can inhibit DNA synthesis in tumor cells, induce cell apoptosis and activate macrophage to produce factors which regulate the function of B, T, as well as NK cell.

Dienogest, is the next choice of progestin drug class. It has high selectivity binding in progesterone receptors, inhibits cytokine secretion in endometriosis stroma cell and induces apoptosis in endometriosis cell. Dienogest also has slight inhibitory effect against estradiol, so it can deminisce the symptoms due to hypoestrogenic such as decresing in bone mass density.

ELIGIBILITY:
Inclusion Criteria:

* female ratus rat type
* having normal estrus cycle

Exclusion Criteria:

* nothing

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — we used female rats to make a model of endometriosis
Enrollment: 120 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
mRNA expressions of Bax, Bcl, Cleaved Caspase 3, IL-1B, and PGE 2 | through study completion, an average of 6 months
  The expression of Bax, Bcl-2, ad Caspase 3, IL-1B, PGE2 mRNA was carried out by isolating the RNA samples of endometriosis tissue based on the modified QIAamp RNA Blod Mini Handbook protocol. RNA spectrophotometric measurments and cDNA synthesis were carried out based on the Instruction Manual ReverTra Ace qPCR RT Master Mix with gDNA Remover protocol (Toyobo 2017: 2). In real-time PCR examination, the melting temperature (Tm) was determined to perform Quantitative Real-time PCR (Q-PCR) based on the QuantiTech SYBR Green PCR Handbook protocol (Qiagen 2011: 11) using a 3-step cycling cycle. The results were then compared with the standard curve and analyzed
Mollecular docking | during the procedure
  Twenty-three compounds contained in Propolis were tested by screening using rule of 5 (Lipinski's rule), screening results determine which compounds can enter the body and can work in endometriosis tissue. Furthermore, the three-dimensional shape is made of compounds which have passed the first stage. This process was created using the Marvin Sketch program. Furthermore, the compound that has been formed is stored as a ligand with extension pdb (protein data bank). Look for NFĸB receptor proteins, estrogen A, estrogen B, progesterone A and progesterone B in the protein data bank, which will be stored as protein. Ligands and proteins are tested using standard Lamarckian algorithms in the Autodock program. The results obtained are in the form of bond energy (ΔG), where smaller results indicate a higher likelihood of interaction
Lession size | during the procedure
  In the second laparotomy (before the treatment are given) the investigators take a picture of the lession (as the beginning lession). Then the investigators give the treatment. After the treatment are done, the investigators do the necropsy to take a picture after the treatment was given to compare it with the beginning
The normality of estrus cycle after the treatment | during the procedure
  Vaginal discharge of the rat obtained through vaginal lavage was fixed using 90% alcohol solution and stained using Giemsa. The specimen was examined microscopically to determined its estrous cycle

SECONDARY OUTCOMES:
Organs morpholgy after the treatment | through study completion, an average of 6 months
  In the necropsy, the investigators take ovarium, uterus, and peritonium to see if there's any change in morphology after the treatment was given

CONTACTS AND LOCATIONS:
Overall Officials: Wachyu Hadisaputra, Prof, dr, SpOG, Principal Investigator — Lecturer at Obgyn Department, Indonesia University
Locations (1):
- Animal Laboratory of Indonesia University, Jakarta, Capital Special Region, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT04374006/Prot_SAP_000.pdf